CLINICAL TRIAL: NCT05266053
Title: Negative Pressure Wound Therapy-PICO: Cosmesis in Repeat C-Sections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lisa Annette Mims, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008549700
Record Dates: First submitted 2022-02-01; First posted 2022-03-04 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hypertrophic Skin Condition of Anterior Abdomen

STUDY DESIGN:
Intervention Model Description: Women will be randomized to placement of a PICO 7 dressing or a standard abdominal dressing at the time of cesarean. The standard abdominal dressing will be removed approximately on postoperative day (POD) 1-2 and the PICO 7 dressing will be removed approximately on POD 3-4 (prior to discharge). If the patient with a PICO dressing remains inpatient for longer than 7 postoperative days, the PICO dressing will be removed prior to POD 7, in accordance with device instructions. Participants in both groups will be sent POSAS surveys at the two, four and six week visit window with primary outcome being aesthetic appearance (cosmesis) at six weeks. Observers (healthcare providers) will complete a POSAS survey at the postpartum visit (~4-6 weeks postoperative) to rate scar quality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): This group will have a PICO negative pressure wound treatment device applied to their surgical wound site.
  Interventions: Device: PICO 7 dressing
- Control Group (Other): Standard Intervention. This group will have a standard wound dressing (gauze, bandage) applied to their surgical wound site.
  Interventions: Other: Standard wound dressing

INTERVENTIONS:
Device: PICO 7 dressing — The PICO 7 dressing consists of a negative pressure wound therapy pump (NPWT) connected to an absorbent gentle adhesive dressing that is applied to a wound. When the pump is activated, it acts by pulling excess fluid from the wound. The dressing absorbs this fluid and helps to prevent bacteria from entering the wound. It has been shown to prevent wound infections and promote healing.
  Arms: Treatment Group
Other: Standard wound dressing — Standard abdominal dressing at the time of cesarean
  Arms: Control Group

SUMMARY:
There are millions of births each year with 32% of women undergoing cesarean sections (C-sections), which results in skin scarring. Repeat C-sections increased by 178% from 1979-2010. Given the frequency of C-sections, it is important to achieve a desirable cosmetic outcome.

The PICO 7 dressing consists of a negative pressure wound therapy pump (NPWT) connected to an absorbent gentle adhesive dressing that is applied to a wound. When the pump is activated, it acts by pulling excess fluid from the wound. The dressing absorbs this fluid and helps to prevent bacteria from entering the wound. It has been shown to prevent wound infections and promote healing. This study aims to compare the aesthetic appearance by using The Patient and Observer Scar Assessment Scale (POSAS) scar assessment scale following closed incision negative pressure therapy with a PICO 7 dressing to the standard abdominal dressing in women undergoing repeat cesarean sections

DETAILED DESCRIPTION:
Single, randomized controlled trial in women undergoing a repeat cesarean delivery. Women will be randomized to placement of a PICO 7 dressing or a standard abdominal dressing at the time of cesarean. The standard abdominal dressing will be removed approximately on postoperative day (POD) 1-2 and the PICO 7 dressing will be removed approximately on POD 3-4 (prior to discharge). If the patient with a PICO dressing remains inpatient for longer than 7 postoperative days, the PICO dressing will be removed prior to POD 7, in accordance with device instructions. Participants in both groups will be sent POSAS surveys at the two, four and six week visit window with primary outcome being aesthetic appearance (cosmesis) at six weeks. Observers (healthcare providers) will complete a POSAS survey at the postpartum visit (~4-6 weeks postoperative) to rate scar quality.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled or non-labor repeat cesarean delivery
* One or more prior cesarean section(s) with prior pfannenstiel incision scar
* Gestational age > 23 weeks
* Age 18 and older

Exclusion Criteria:

* Patients with malignancy in the wound bed or margins of the wound
* Non-enteric and unexplored fistulas
* Necrotic tissue with eschar present
* Exposed arteries, veins, nerves or organs
* Exposed anastomotic sites
* Cellulitis or evidence of active infection
* Known allergy to adhesive tape
* Patient unwilling to follow-up
* Contraindication to NPWT

  * Bleeding disorder
  * Therapeutic anticoagulation
  * Allergy to any component of the dressing (perhaps list these as you will need to know to confirm eligibility of each patient)
  * Prior irradiated skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant transgender males may participate in the study.
Enrollment: 24 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mims, MD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown BC, Moss TP, McGrouther DA, Bayat A. Skin scar preconceptions must be challenged: importance of self-perception in skin scarring. J Plast Reconstr Aesthet Surg. 2010 Jun;63(6):1022-9. doi: 10.1016/j.bjps.2009.03.019. Epub 2009 Jun 5. PMID 19501559
- [Background] Figueroa D, Jauk VC, Szychowski JM, Garner R, Biggio JR, Andrews WW, Hauth J, Tita AT. Surgical staples compared with subcuticular suture for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Jan;121(1):33-8. doi: 10.1097/aog.0b013e31827a072c. PMID 23262925
- [Background] Hyldig N, Birke-Sorensen H, Kruse M, Vinter C, Joergensen JS, Sorensen JA, Mogensen O, Lamont RF, Bille C. Meta-analysis of negative-pressure wound therapy for closed surgical incisions. Br J Surg. 2016 Apr;103(5):477-86. doi: 10.1002/bjs.10084. PMID 26994715
- [Background] Hyldig N, Vinter CA, Kruse M, Mogensen O, Bille C, Sorensen JA, Lamont RF, Wu C, Heidemann LN, Ibsen MH, Laursen JB, Ovesen PG, Rorbye C, Tanvig M, Joergensen JS. Prophylactic incisional negative pressure wound therapy reduces the risk of surgical site infection after caesarean section in obese women: a pragmatic randomised clinical trial. BJOG. 2019 Apr;126(5):628-635. doi: 10.1111/1471-0528.15413. Epub 2018 Sep 7. PMID 30066454
- [Background] Ekin M, Dagdeviren H, Caypinar SS, Erdogan B, Ayag ME, Cengiz H, Yasar L, Helvacioglu C. Comparative cosmetic outcome of surgical incisions created by the PEAK Plasma Blade and a scalpel after cesarean section by Patient and Observer Assessment Scale (POSAS): A randomized double blind study. Taiwan J Obstet Gynecol. 2018 Feb;57(1):68-70. doi: 10.1016/j.tjog.2017.12.011. PMID 29458906
- [Background] Truong PT, Lee JC, Soer B, Gaul CA, Olivotto IA. Reliability and validity testing of the Patient and Observer Scar Assessment Scale in evaluating linear scars after breast cancer surgery. Plast Reconstr Surg. 2007 Feb;119(2):487-94. doi: 10.1097/01.prs.0000252949.77525.bc. PMID 17230080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from medical clinic and in-patient admissions.
Pre-assignment Details: There are no pre-assignment factors that impact participant enrollment.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 12 | 12
Completed | 4 | 8
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 12 | 12 | 24
  Sex: Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Scar Assessment [Median (Full Range); unit: units on a scale] — Patients were evaluated using the Patient and Observer Scar Assessment (POSAS) Scale.
  Patient is asked as series of subjective questions regarding pain, color, stiffness, thickness, irregularity, itching, and overall impression. Participants respond with a scale of 1 - 10 with 10 as the most severe appearance and 1 as the least severe appearance. These scores are summed for a total value of 6 (total best outcome) through 60 (total worst outcome).
  The full range provided reflects the actual collected data from the participants. Population: Subjects analyzed were much lower due to lack of patient response and patients loss to follow up.
  units on a scale
    number analyzed (Participants) | 5 | 2 | 7
    (all) | 19 [16 to 32] | 33 [17 to 49] | 26 [16 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Subjective Cosmetic Result
Description: Patients were evaluated using the Patient and Observer Scar Assessment (POSAS) Scale.
  Patient is asked as series of subjective questions regarding (vascularity, pigmentation, thickness, relief, pliability, surface area). Participants respond with a scale of 1 - 10 with 10 as the most severe appearance and 1 as the least severe appearance. These scores are summed for a total value of 6 (total best outcome) through 60 (total worst outcome).
  The full range provided reflects the actual collected data from the participants.
Time Frame: Week 6
Population: The only subjects analyzed were those that were evaluated in week 6
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 8 | 4
units on a scale | 13 [10 to 16.5] | 26.5 [16 to 36.5]

2. Primary Outcome: Patient Satisfaction With Wound Appearance
Description: Scale of 1 - 10 with 1 being least satisfied and 10 being most satisfied
Time Frame: Week 6
Population: Some participants did not complete surveys so the Overall Number of Participants reflects participants with scale data collected.
  The full range provided reflects the actual collected data from the participants.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale | 2 [2 to 2] | 7 [4 to 10]

3. Secondary Outcome: Procedure Time in Minutes
Description: Procedure time in minutes
Time Frame: Start of surgery until application of wound vac immediately post-procedure
Population: Data was not collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Analog Pain Scores 48 Hours
Description: Participants respond with a scale of 1 - 10 with 10 as most severe and 1 as not at all.
  The full range provided reflects the actual collected data from the participants.
Time Frame: 48 hours after surgery
Population: No data was collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Analog Pain Scores 72 Hours
Description: Participants respond with a scale of 1 - 10 with 10 as the most severe and 1 being no pain at all.
  The full range provided reflects the actual collected data from the participants.
Time Frame: 72 hours after surgery
Population: No Data was collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Analog Pain Scores @4 Weeks
Description: as for outcome 5
Time Frame: 4 weeks after surgery at postpartum visit
Population: Some participants did not complete surveys so the Overall Number of Participants reflects participants with scale data collected.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 2
score on a scale | 2 [1 to 5] | 6 [2 to 10]

7. Secondary Outcome: Analog Pain Scores @6 Weeks
Description: as for outcome 5
Time Frame: 6 weeks after surgery at postpartum visit
Population: as for outcome 6
Measure: Median (Full Range); unit: score on a scale
Groups:
- Treatment: This group will have a PICO negative pressure wound treatment device applied to their surgical wound site.
  PICO 7 dressing: The PICO 7 dressing consists of a negative pressure wound therapy pump (NPWT) connected to an absorbent gentle adhesive dressing that is applied to a wound. When the pump is activated, it acts by pulling excess fluid from the wound. The dressing absorbs this fluid and helps to prevent bacteria from entering the wound. It has been shown to prevent wound infections and promote healing.
- Control: Standard Intervention. This group will have a standard wound dressing (gauze, bandage) applied to their surgical wound site.
  Standard wound dressing: Standard abdominal dressing at the time of cesarean
Arm/Group | Treatment | Control
Number analyzed (Participants) | 8 | 4
score on a scale | 1.5 [1 to 3] | 1.5 [1 to 4]

8. Secondary Outcome: Incision Healing Complications up to 42 Days Postoperatively
Description: Number of Participants with Incision Healing Complications up to 42 Days Postoperatively
Time Frame: 42 day after surgery
Population: Some participants did not complete follow up as scheduled. Data analysed reflects participants with collected data.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: This group will have a PICO negative pressure wound treatment device applied to their surgical wound site.
  PICO 7 dressing: The PICO 7 dressing consists of a negative pressure wound therapy pump (NPWT) connected to an absorbent gentle adhesive dressing that is applied to a wound. When the pump is activated, it acts by pulling excess fluid from the wound. The dressing absorbs this fluid and helps to prevent bacteria from entering the wound. It has been shown to prevent wound infections and promote healing.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 8 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Lack of self guided patient participation or return of survey request.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT05266053/Prot_003.pdf
  • Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT05266053/SAP_001.pdf
  • Informed Consent Form (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT05266053/ICF_004.pdf